CLINICAL TRIAL: NCT06751173
Title: Effects of Static Core Stability Versus Extension Exercises Program on Pain, Range of Motion, and Functional Disability in Patients With Chronic Low Back Pain
Brief Title: Static Core Stability vs. Extension Exercises for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Maryam Arshad
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Chronic Low-back Pain (cLBP)
Keywords: Low back pain; core stability; strengthing
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The Group A will be treated with Static Core Stability exercises and common treatment.
  i. Plank: Press the hands and knees to the floor with the back in a neutral position and wrists aligned directly under the shoulders.
  ii. Side Plank: Lie on the side with knees bent and prop the upper body up on the elbow.
  iii. Shoulder Bridge: Raise the pelvis off the floor until only the head, neck, shoulders, and feet are touching the mat. Place the hands at the waist.
  iv. Static Crunch: Lie on the back with the feet flat on the floor and the knees bent at a 90-degree angle.
  v. Leg Lift: Lie straight on the floor, keep the arms at the sides, and slowly lift both legs into the air.
  Interventions: Other: Static Core Stability exercises; Other: Spinal Mobilization
- Group B (Active Comparator): The second group will consist of McKenzie exercises with common treatment.
  i. Prone Extension (Positioned): Lie on the stomach with pillows placed under the chest for comfort.
  ii. Prone Extension on Elbow: Keep the back and buttocks relaxed and rise up on the elbows as high as possible.
  iii. Prone Press-ups: Place the hands beside the shoulders. Keep the back and buttocks relaxed, and use the arms to press up.
  iv. Standing Extension: Stand with feet apart and hands on the small of the back with fingers pointing backward. Bend backward at the waist while supporting the trunk with the hands.
  v. Sideglide in Standing: Stand at a right angle to the wall about 2 feet away. Lean the shoulder into the wall.
  Common Treatment: Spinal mobilization with central-unilateral posterior-anterior and lateral glide.
  Interventions: Other: Mckenzie exercises; Other: Spinal Mobilization

INTERVENTIONS:
Other: Static Core Stability exercises — i. Plank: Press the hands and knees to the floor with the back in a neutral position and wrists aligned directly under the shoulders.
  ii. Side Plank: Lie on the side with knees bent and prop the upper body up on the elbow.
  iii. Shoulder Bridge: Raise the pelvis off the floor until only the head, neck, shoulders, and feet are touching the mat. Place the hands at the waist.
  iv. Static Crunch: Lie on the back with feet flat on the floor and knees bent at a 90-degree angle.
  v. Leg Lift: Lie straight on the floor, keep the arms at the sides, and slowly lift both legs into the air.
  Arms: Group A
Other: Mckenzie exercises — i. Prone Extension (Positioned): Lie on the stomach with pillows placed under the chest for comfort.
  ii. Prone Extension on Elbow: Keep the back and buttocks relaxed and rise up on the elbows as high as possible.
  iii. Prone Press-ups: Place the hands beside the shoulders. Keep the back and buttocks relaxed, and use the arms to press up.
  iv. Standing Extension: Stand with feet apart and hands on the small of the back with fingers pointing backward. Bend backward at the waist, supporting the trunk with the hands.
  v. Side glide in Standing: Stand at a right angle to the wall about 2 feet away. Lean the shoulder into the wall.
  Arms: Group B
Other: Spinal Mobilization — Central-Unilateral posterio anterior and lateral glide

SUMMARY:
Chronic back pain is posteriorly occurring multi-causes pain that most commonly occurred due to lumber strains and sprains. It usually lasts 12 weeks (03 months) or longer. It is exacerbated by prolonged sitting, lifting heavy weights and sudden awkward movements. The aim of study will be to compare the effects of static core stability versus extension exercises program on pain, range of motion and functional disability in patients with chronic low back pain. A Randomized Clinical Trial will be conducted at Riphah Clinic Lahore and Jinnah Hospital Lahore through lottery methode technique on 30 patients which will be allocated using simple random sampling through sealed opaque enveloped into Group A and Group B. Group A will be treated with static core stabilization exercises and Group B will be treated with lumber extension exercises at the frequency of 2 sets with 10 repetitions and thrice a week. Outcome measures will be conducted through pain, range of motion and functional disability questionnaire after 6 weeks. Data will be analyzed during SPSS software version 21. After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

DETAILED DESCRIPTION:
Low back pain is defined as pain and discomfort at costal margins and lower gluteal folds that does not radiate in lower limbs and also not attributed to any specific disease(1). Globally, more than half a billion people are suffering from Chronic Low Back pain which results in poor Quality of life (QOL) among people(2) and indirect costs (work absenteeism, productivity loss) account for more than half of the total costs.Although most patients with acute LBP show rapid improvements in pain and disability within 1 month,(3) between 4% and 25% of patients drift to chronicity. The prevalence of chronic low back pain (CLBP) increases linearly from the third decade of life until the age of 60 years, with CLBP being more prevalent in women.(4) When LBP persists for 12 weeks or longer,we say it as chronic low back pain(5). Chronic low back pain can cause fatigue, noctural pain hence interrupting sleep,depressed mood and ADLs limitations.There are a number of factors identified which may lead to LBP including stress, incorrect posture, awkward sleeping position, weight gains, gender, age, prolonged sitting time, family history, history of fall/trauma, and socioeconomic status. A sedentary lifestyle has a major role in developing LBP(2). The word Core is a word derived from English, which is used to mean seed. It is the midpoint of the body, where the center of gravity of the human body lay. It includes your pelvis, lower back, hips and stomach.Globally accepted definition of core stability is ""Comprises of the lumbopelvic-hip complex and is the capacity to maintain the equilibrium of the vertebral column within its physiologic limits by reducing displacement from perturbations and maintaining structural integrity."(6)(7)(8)(9)(10). The body's core region is sometimes referred to as the torso or the trunk. The major muscles involved in core stability include the pelvic floor muscles, transversus abdominis, multifidus, internal and external obliques, rectus abdominis, erector spinae (sacrospinalis) especially the longissimus thoracis, and diaphragm. Core stability has a high established reliability in improving the trunk muscle performance as core muscles supporting the lumbo-pelvic-hip complex, researchers have reported that core stability training could improve not only trunk function but also balance and mobility(11). It also consist of movements that increase the flexibility and strength of the body also increases muscle endurance and cardiovascular fitness levels. They develop psychomotor skills and coordination.(13). In static core exercises, such as the standard plank, side plank, and lifted leg/arm planks, the joint and muscle either work against an immovable force or is held in a static position with some resistance.(12)Majewski-Schrage et al. state that core stability has overcome the physical health approach over time, becoming a part of health and physical performance issues with different approaches, and according to them, this situation is now 4 related to physical fitness, rehabilitation programs, back-spine problems, and performance(13). Lumbar extension is the bending backward of the spine.Back extension is one of the most needed motions of the spine to improve posture and to keep balance within the body.Back extension exercises (sometimes also called hyperextensions) can strengthen lower back muscles and work by centralizing pain.Acording to Brett Sears, PT's article Lumbar Extension and How It Helps Back Pain published on march 2023 stated as 'Lumbar extension exercises are used to increase range of motion (ROM) in people with lower back pain. Lumbar extension places stress and pressure on the backside of your intervertebral discs, those soft, squishy shock absorbers in your spine." Back extension exercises specifically focus on the low back and the erector spinae muscle group (form the intermediate layer of the back muscles and comprise three subgroup) which help to support, protect, and extend your lower spinal column and entire back. Back extension muscles may also include the middle and upper back muscles as well as the oblique muscles for stabilization(14).In this research we will focus on pelvic tilt, cobra lift, cat and camel stretch, partial curl and gluteal stretch back extension exercises. To the best of our knowledge, there is no study that has so far evaluated the clinical outcome of static core stabilization versus back extension exercises with lumber mobilization as common treatment. In this current study, we will analyze and will be able to identify the most effective intervention between static core stability and back extension exercises on patients with chronic low back pain. Furthermore, we will evalute results on basis of effects on pain intensity, range of motion and functional disability within patients of both groups.

ELIGIBILITY:
INCLUSION CRITERIA:

* Minimum 03 months of chronicity of low back pain.
* No radiating leg pain.
* Moderate pain (NPRS: 3-7)
* Disability score of 19% or greater as evident from the modified Oswestry Disability Questionnaire (MODQ)
* Positive prone instability test

EXCLUSION CRITERIA:

* Chronic systemic boney and soft tissue.
* Recent history of trauma.
* Degenerative joint diseases
* Psychiatric diseases.
* Ongoing radiotherapy, chemotherapy and steroid therapy.
* Localized infection in lumbar region.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Numeric pain rate scale (NPRS) | baseline, 8 weeks
  The patient's level of pain will be assessed using this scale. The 11-point numeric scale ranges from '0,' representing one pain extreme (e.g., "no pain"), to '10,' representing the other pain extreme (e.g., "pain as bad as can be imagined" or "worst pain imaginable").
Osvestry Disability index (ODI) | baseline, 8 weeks
  This questionnaire will be used to assess disability. The Oswestry Disability Index (ODI) consists of 10 questions completed by the patient, with response options presented as 6-point Likert scales. Scores range from 0% (no disability) to 100% (most severe disability).
Inclinometer | baseline, 8 weeks
  The range of motion of the lower back will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Arshad, DPT, Principal Investigator — Riphah International University, Lahore
Locations (1):
- Riphah Rehab Training and Research Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No